CLINICAL TRIAL: NCT03270345
Title: Multicentre International One-Day Prevalence Study on Pressure Injuries in Intensive Care Units
Brief Title: One-Day Prevalence Study on Pressure Injuries in Intensive Care Units
Acronym: DecubICUs
Status: Completed | Type: Observational
Sponsor: European Society of Intensive Care Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: DecubICUs
Record Dates: First submitted 2017-08-29; First posted 2017-09-01 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Pressure Injury
Keywords: Decubitus; Pressure; Ulcer; Injuries; Sores; Intensive care
MeSH Terms: conditions — Pressure Ulcer; Ulcer; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to provide an up-to-date, global picture of the extent and patterns of pressure injuries in ICUs. Point prevalence studies are only of value when performed on a vast scale. To sample a representative cohort, it is the intention to recruit about 1200 ICUs with all continents covered and as many countries as possible within each continent.

DETAILED DESCRIPTION:
The objective is to provide an up-to-date, international "global" picture of the extent and patterns of pressure injuries in ICUs. Thereto , the plan is to perform a 1-day, prospective, multicenter point-prevalence study. The large scale of the project should allow thorough epidemiological analyses. More precisely the study will enable to identify:

* major risk factors for pressure ulcer development;
* preventive measures used in distinct ICU populations and countries;
* shortages in the availability of evidence-based measures to prevent pressure sores;
* malpractice pressure sore prevention in particular regions or countries;
* occurrence rates of pressure ulcers with/without accurate adjustment for risk profile and preventive measures taken;
* benchmarking between regions/countries; clinical outcomes associated with pressure ulcers (major organ derangements and mortality);
* economic outcomes associated with pressure ulcers (length of ICU stay) and linking these outcomes with local practice regarding prevention measures applied/available.
* country and regional differences in prevalence of pressure ulcers and outcome.

Pressures ulcer stages will be graded following the classification system jointly developed by the National Pressure Ulcer Advisory Panel and European Pressure Ulcer Advisory Panel.

Data to be recorded include patient demographics, data on severity of underlying disease and acute illness, organ failure, pressure ulcers, major risk factors for pressure ulcers, and measures taken to prevent pressure ulcers.

Statistical Plan

Power Calculation. For a risk factor with a prevalence in the study cohort of only 10% (for example patients with a BMI<20) and an outcome difference of only 5% to be statistically significant(15% vs. 20% in decubitus occurrence rate), a sample size of 5255 patients is required (478 patients with the index risk factor and 4777 without) (alpha=0.05; Beta>0.80).

Data cleaning &missing data. Exceptional values will be traced through distribution plotting. In case of uncertainties, the individual investigators will be contacted. Missing data will be handled by imputation (1, 2). Data quality checks will be performed, such as checks on completeness, consistency, correctness, and uniqueness.

Descriptives. A single final analysis is planned at the end of the study; no interim analyses are planned. Socio-demographic study cohort characteristics will be described as proportions for categorical variables and for continuous variables as mean and standard deviation if normally distributed or median and inter-quartile range if not normally distributed (according to the Kolmogorov-Smirnov test for normality).

The proportion of patients with decubitus (percentage, %, and their 95% confidence intervals) will be reported overall and according to geographic region (continent), country classification by income as defined by The World Bank (high-, upper-middle-, lower-middle-, and low-income countries), percentage of the gross domestic product spent on healthcare (obtained from the World Health Organization), and according to theEducation and Health Human Development Report of the United Nations Development Program. Subsequently, potentialdifferences in prevalence might offer the opportunity to evaluate variances in prevention measures on a large scale.

Modelling. Covariates that will be evaluated on their relationship with the presence of decubitus encompass various organizational aspects of the ICU (e.g. nurse-to-patient ratio), decubitus prevention measures (e.g. type of matrasses used), and patient-specific characteristics (e.g. age, underlying conditions, severity of acute illness, body morphology, BMI,length of ICU stay etc.). Covariates will be considered for adjusted analysis when they have an association with pressure injuries at a statistical level <0.25 in unadjusted (univariate) analysis or because of their clinical relevance. A stepwise approach willbe used to eliminate terms from the regression model; p<0.15 or p<0.10 will beset as the limit to keep covariates in the model.

Relationships with binary outcome variables (e.g. decubitus, mortality) will be assessed by means of unadjusted statistical tests and multivariate logistic regression. The value of additional propensity score correction in the regression model will be assessed. Multinomial logistic regression will be performed to assess independent relationships with decubitus stages. Likewise, linear mixed-effect modelling will be used to assess unadjusted and adjusted relationships with continuous outcome variables (e.g. length of ICU stay and length of hospitalization). Results of logistic regression will be reported as adjusted odds ratios with 95% confidence intervals.

To develop a decubitus prediction model for distinct ICU populations (e.g., trauma, surgical or medical patients) models will be build using machine learning techniques (e.g. Random Forest, Gradient Boosting Machine). In the process different techniques will be applied in order to receive the optimal accuracy. In order to gain insight in the correlation between predictors and variables, regression techniques will be applied, as state above.

For validation of our models the study cohort will be split into a training, test and validation set. As such this gives a fair interpretation of the results. Alternatively ten-fold cross-validation can be applied to prevent overfitting.

Benchmarking for individual centers based on decubitus will be performed by providing directly or indirectly standardized risks based on fixed center effects in a logistic regression model (3, 4). Besides the presence of the binary quality outcome (i.e. decubitus) and the center code, this model also includes patient-specific baseline co-variates to adjust for differential case-mix. The Firth correction will be applied to the logistic regression model to maintain convergence in the presence of very small centers (5).

Statistical analysis will be performed using SPSS and R. The head investigator (SB) is responsible for all statistical analysis. Advanced statistical methods will be executed byMiekeDeschepper (Strategic Policy Cell at Ghent University Hospital).

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (>18 years of age) present on the date of data collection

Exclusion Criteria:

* There are no exclusion criteria. All patients should be included. Patients with severe clinical conditions not allowing safe pressure ulcer identification should not be evaluated for the respective risk zones. If it is known that the patient has a pressure ulcer at the body sites that cannot be safely evaluated, the stage of the pressure ulcer should be recorded as previously known. If it is unknown whether the patient has a pressure ulcer at these body sites, this should be indicated with a '?' in the Case Report Form

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All , adult ICU patients present in the ICU.
Sampling Method: Non-Probability Sample
Enrollment: 13340 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
major risk factors for pressure injury development. | on the data collection day of 18 May 2018 (84 days follow-up)
  Pressures injury stages will be graded following the classification system jointly developed by the National Pressure Ulcer Advisory Panel, European Pressure Ulcer Advisory Panel, and Pan Pacific Pressure Injury Alliance. Data to be recorded include patient demographics, data on severity of underlying disease and acute illness, organ failure, pressure ulcers, major risk factors for pressure ulcers, and measures taken to prevent pressure injuries.

CONTACTS AND LOCATIONS:
Overall Officials: Stijn BLOT, Principal Investigator — Full Professor, Dept. of Internal Medicine, Faculty of Medicine & Health Science, Ghent University, Belgium; Sonia LABEAU, Principal Investigator — Lecturer at University College Ghent, Belgium
Locations (1):
- All Centers From All Over the World Willing to Contribute Are Welcome, Brussels, Belgium

REFERENCES:
- [Background] Bennett G, Dealey C, Posnett J. The cost of pressure ulcers in the UK. Age Ageing. 2004 May;33(3):230-5. doi: 10.1093/ageing/afh086. PMID 15082426
- [Background] Keller BP, Wille J, van Ramshorst B, van der Werken C. Pressure ulcers in intensive care patients: a review of risks and prevention. Intensive Care Med. 2002 Oct;28(10):1379-88. doi: 10.1007/s00134-002-1487-z. Epub 2002 Sep 7. PMID 12373461
- [Background] Blot S, Cankurtaran M, Petrovic M, Vandijck D, Lizy C, Decruyenaere J, Danneels C, Vandewoude K, Piette A, Vershraegen G, Van Den Noortgate N, Peleman R, Vogelaers D. Epidemiology and outcome of nosocomial bloodstream infection in elderly critically ill patients: a comparison between middle-aged, old, and very old patients. Crit Care Med. 2009 May;37(5):1634-41. doi: 10.1097/CCM.0b013e31819da98e. PMID 19325489
- [Background] Iranmanesh S, Rafiei H, Sabzevari S. Relationship between Braden scale score and pressure ulcer development in patients admitted in trauma intensive care unit. Int Wound J. 2012 Jun;9(3):248-52. doi: 10.1111/j.1742-481X.2011.00852.x. Epub 2011 Sep 13. PMID 21910830
- [Background] Manzano F, Navarro MJ, Roldan D, Moral MA, Leyva I, Guerrero C, Sanchez MA, Colmenero M, Fernandez-Mondejar E; Granada UPP Group. Pressure ulcer incidence and risk factors in ventilated intensive care patients. J Crit Care. 2010 Sep;25(3):469-76. doi: 10.1016/j.jcrc.2009.09.002. Epub 2009 Oct 30. PMID 19879730
- [Background] Nijs N, Toppets A, Defloor T, Bernaerts K, Milisen K, Van Den Berghe G. Incidence and risk factors for pressure ulcers in the intensive care unit. J Clin Nurs. 2009 May;18(9):1258-66. doi: 10.1111/j.1365-2702.2008.02554.x. Epub 2008 Dec 11. PMID 19077028
- [Background] Terekeci H, Kucukardali Y, Top C, Onem Y, Celik S, Oktenli C. Risk assessment study of the pressure ulcers in intensive care unit patients. Eur J Intern Med. 2009 Jul;20(4):394-7. doi: 10.1016/j.ejim.2008.11.001. Epub 2008 Dec 6. PMID 19524181
- [Background] Harvey SE, Parrott F, Harrison DA, Bear DE, Segaran E, Beale R, Bellingan G, Leonard R, Mythen MG, Rowan KM; CALORIES Trial Investigators. Trial of the route of early nutritional support in critically ill adults. N Engl J Med. 2014 Oct 30;371(18):1673-84. doi: 10.1056/NEJMoa1409860. Epub 2014 Oct 1. PMID 25271389
- [Background] Matos LS, Duarte NLV, Minetto RdCs, (2010) Incidence and prevalence of ulcer for pressure in CTI of a Public Hospital of DF. Revista Eletronica de Enfermagem 12: 719-726
- [Background] European Pressure Ulcer Advisory Panel and National Pressure Ulcer Advisory Panel (2009) Prevention and treatment of pressure ulcers: quick reference guide. National Pressure Ulcer Advisory Panel, Washington DC
- [Background] Schafer JL. Multiple imputation: a primer. Stat Methods Med Res. 1999 Mar;8(1):3-15. doi: 10.1177/096228029900800102. PMID 10347857
- [Background] Schafer JL, Olsen MK. Multiple Imputation for Multivariate Missing-Data Problems: A Data Analyst's Perspective. Multivariate Behav Res. 1998 Oct 1;33(4):545-71. doi: 10.1207/s15327906mbr3304_5. PMID 26753828
- [Background] Van Messem M, Varewyck M: Evaluating hospital peformance Risk Standard package. Ghent: Ghent University; 2015
- [Background] Varewyck M, Vansteelandt S, Eriksson M, Goetghebeur E. On the practice of ignoring center-patient interactions in evaluating hospital performance. Stat Med. 2016 Jan 30;35(2):227-38. doi: 10.1002/sim.6634. Epub 2015 Aug 24. PMID 26303843
- [Background] Firth D: Bias Reduction of Maximum Likelihood Estimates.Biometrika Vol. 80, No. 1 (Mar., 1993), pp. 27-38
- [Derived] Dejonckheere M, Antonelli M, Arvaniti K, Blot K, CreaghBrown B, de Lange DW, De Waele J, Deschepper M, Dikmen Y, Dimopoulos G, Eckmann C, Francois G, Girardis M, Koulenti D, Labeau S, Lipman J, Lipovestky F, Maseda E, Montravers P, Mikstacki A, Paiva J, Pereyra C, Rello J, Timsit J, Vogelaers D, Blot S; Abdominal Sepsis Study (AbSeS) group on behalf of the Trials Group of the European Society of Intensive Care Medicine. Epidemiology and risk factors for mortality in critically ill patients with pancreatic infection. J Intensive Med. 2023 Aug 30;4(1):81-93. doi: 10.1016/j.jointm.2023.06.004. eCollection 2024 Jan. PMID 38263964
- [Derived] Rubulotta F, Brett S, Boulanger C, Blackwood B, Deschepper M, Labeau SO, Blot S; UK Collaborating Site Investigators; DecubICUs study team and the European Society of Intensive Care Medicine Trials' Group UK Collaborators. Prevalence of skin pressure injury in critical care patients in the UK: results of a single-day point prevalence evaluation in adult critically ill patients. BMJ Open. 2022 Nov 23;12(11):e057010. doi: 10.1136/bmjopen-2021-057010. PMID 36418122
- [Derived] De Pascale G, Antonelli M, Deschepper M, Arvaniti K, Blot K, Brown BC, de Lange D, De Waele J, Dikmen Y, Dimopoulos G, Eckmann C, Francois G, Girardis M, Koulenti D, Labeau S, Lipman J, Lipovetsky F, Maseda E, Montravers P, Mikstacki A, Paiva JA, Pereyra C, Rello J, Timsit JF, Vogelaers D, Blot S; Abdominal Sepsis Study (AbSeS) group and the Trials Group of the European Society of Intensive Care Medicine. Poor timing and failure of source control are risk factors for mortality in critically ill patients with secondary peritonitis. Intensive Care Med. 2022 Nov;48(11):1593-1606. doi: 10.1007/s00134-022-06883-y. Epub 2022 Sep 23. PMID 36151335
- [Derived] Arvaniti K, Dimopoulos G, Antonelli M, Blot K, Creagh-Brown B, Deschepper M, de Lange D, De Waele J, Dikmen Y, Eckmann C, Einav S, Francois G, Fjeldsoee-Nielsen H, Girardis M, Jovanovic B, Lindner M, Koulenti D, Labeau S, Lipman J, Lipovestky F, Makikado LDU, Maseda E, Mikstacki A, Montravers P, Paiva JA, Pereyra C, Rello J, Timsit JF, Tomescu D, Vogelaers D, Blot S; Abdominal Sepsis Study (AbSeS) Group on behalf of the Trials Group of the European Society of Intensive Care Medicine. Epidemiology and age-related mortality in critically ill patients with intra-abdominal infection or sepsis: an international cohort study. Int J Antimicrob Agents. 2022 Jul;60(1):106591. doi: 10.1016/j.ijantimicag.2022.106591. Epub 2022 Apr 20. PMID 35460850